CLINICAL TRIAL: NCT00324753
Title: Improving Patient-Provider Communication For Colorectal Cancer Screening
Brief Title: Quality Improvement of Patient-Provider Communication For Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIR 03-252
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
Keywords: cancer; screening; communication; prevention
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Communication | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Communication sheet
  Interventions: Behavioral: Communication
- Control (Other): Standard of care brochures
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Communication — Communication sheet
  Arms: Intervention
Behavioral: Standard of care — Standard of care brochures
  Arms: Control

SUMMARY:
The immediate objective of this proposal is to assess the effectiveness of a multi-faceted intervention to improve patient-provider communication about colorectal cancer screening in improving patient adherence with colorectal cancer screening recommendations. This intervention consists of: (1) guiding the communication process through patient activation to initiate a colorectal cancer screening discussion; (2) optimizing communication content through the use of a prompt sheet; and (3) cueing the provider to assess patient perception of the communication. The long-term objective of our research program is to maximize colorectal cancer screening rates throughout the VA through widespread adoption of clinically feasible approaches to enhance patient-provider communication.

DETAILED DESCRIPTION:
In the United States, colorectal cancer is the third most common cancer and the second leading cause of cancer mortality with over 56,000 deaths in 2004). Early detection through screening decreases the mortality associated with the disease. However, adherence with current screening recommendations is low. A survey of the general population indicates that only 53.1% of Americans, age 50 years and older for whom colorectal cancer screening is recommended, are up-to-date with this preventive service. While colorectal cancer screening rates with the VA Healthcare System (VHA) are better than in the general population (75% in Fiscal Year (FY) 2005), they are lower than performance rates for other types of cancer screening (e.g., mammography) in VHA. Further, numerous VA medical centers report colorectal cancer screening rates below the level considered satisfactory.

ELIGIBILITY:
Inclusion Criteria:

Provider Eligibility:

* Primary care providers (MD, Certified Registered Nurse Practitioner (CRNP), or PA) at the study sites who see patients in the primary care setting at least 1 day per week and had no involvement in the design of the study are eligible for enrollment in the study.

Patient Eligibility:

* Primary care patients who are not "up-to-date" with colorectal cancer screening are the targeted population for study enrollment.
* Up-to-date with colorectal cancer screening is defined as having completed one of the following:

  * fecal occult blood testing within the past year
  * sigmoidoscopy within the past 5 years
  * colonoscopy within the past 10 years
  * barium enema within the past 5 years.
* Other patient eligibility criteria are:

  * Primary Care Provider (PCP) enrolled in the study
  * clinic visit scheduled with the enrolled PCP during the recruitment period
  * English speaking
  * no prior history of colorectal cancer or adenomatous polyps
  * no prior history of inflammatory bowel disease

Exclusion Criteria:

* Patients who are deemed clinically not appropriate for colorectal cancer screening due to severe comorbidity and/or limited life expectancy as determined by the patient's primary care provider will be excluded from the study.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce S. Ling, MD MPH, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ling BS, Trauth JM, Fine MJ, Mor MK, Resnick A, Braddock CH, Bereknyei S, Weissfeld JL, Schoen RE, Ricci EM, Whittle J. Informed decision-making and colorectal cancer screening: is it occurring in primary care? Med Care. 2008 Sep;46(9 Suppl 1):S23-9. doi: 10.1097/MLR.0b013e31817dc496. PMID 18725829
- See also: Click here for more information about this study: Improving Patient-Provider Communication For Colorectal Cancer Screening — http://www.pittsburgh.va.gov/docs/quics_booklet.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Intervention arm- Prompting by prevention nurses and a communication sheet provided
  A prevention nurse addressed the process of communication by activating the patient to initiate and conduct a discussion on colorectal cancer screening at the clinical encounter with their PCP. The prevention nurse also provided a talking guide to the patient which was a double-sided single sheet that contained specific communication content pertinent to colorectal cancer screening that should be addressed with the PCP during the clinical encounter and included specific information on fecal occult blood testing and colonoscopy. The patient and PCP could determine the depth at which the communication occurred depending on factors such as time and competing clinical demands. Included in this talking guide were items designed to assist the PCP in assessing the patient's perception of the communication that occurred during the clinical encounter.
- Control: Usual care arm which consisted of standard of care brochures available clinically. No communication prompts or guides provided for those in Arm 2.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 190 | 264
Completed | 190 | 264
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 190 | 264 | 454
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 50-59 | 114 | 160 | 274
  Age (years): 60-69 | 67 | 96 | 163
  Age (years): 70 and older | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 22 | 59
  Male | 153 | 242 | 395
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 172 | 241 | 413
  Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 68 | 82 | 150
  Race: African American | 103 | 166 | 269
  Race: Other | 14 | 9 | 23
  Race: Not Answered | 5 | 7 | 12
Charlson Comorbidity Index [Count of Participants; unit: Participants] — The Charlson Comorbidity Index is a measure of comorbid burden. The index is a weighted sum of the presence of up to 22 comorbid conditions, which are each provided a weight of 1, 2, 3, or 6 as originally derived based on the contribution of each comorbid condition to one-year mortality. A score of 0, indicates the absence of the measured comorbidities, and higher scores indicate a higher level of comorbid burden, with a higher predicted risk of death.
  Participants
    0 | 75 | 137 | 212
    1 | 62 | 61 | 123
    2 or more | 53 | 66 | 119
Family History of Colorectal Cancer or Polyps [Count of Participants; unit: Participants]
  History of Colorectal Cancer | 20 | 26 | 46
  History of Polyps only | 16 | 18 | 34
  History of Neither | 154 | 220 | 374
Education [Count of Participants; unit: Participants]
  < High School Graduate | 16 | 160 | 176
  High School Graduate | 52 | 96 | 148
  Post High School | 120 | 8 | 128
  Not Answered | 2 | 0 | 2
Site [Count of Participants; unit: Participants]
  Chicago | 72 | 116 | 188
  Houston | 49 | 61 | 110
  Pittsburgh | 69 | 87 | 156

OUTCOME MEASURES:

1. Primary Outcome: Completion of Colorectal Cancer Screening Tests
Description: A survey collected data on patient demographic characteristics, family history of colorectal cancer or polyp, and provider recommendation for colorectal cancer screening, if any. In addition, we asked patients whether colorectal cancer screening was discussed at the visit. If the response was yes, we then asked patients how satisfied they were with the PCP communication during the visit in general using a 5-point Likert scale to a number of items describing the communication. A medical record review was conducted to collect data on provider ordering and patient completion of the following colorectal cancer screening tests during the study period (i.e., 6 months from the time of the clinical encounter): fecal occult blood testing, sigmoidoscopy, or colonoscopy.
Time Frame: 6-12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 190 | 264
Participants
  CRC Test Completed | 102 | 142
  CRC Test Not Completed | 88 | 122
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .005, Mixed Models Analysis — p-value based on a test of any treatment difference by site; The model was run using the xtlogit command in Stata and was adjusted for all of the reported baseline characteristics

2. Primary Outcome: Quality of Communication
Description: Patient satisfaction with the discussion of Colorectal Cancer (CRC) screening with the primary care provider (PCP).
Time Frame: immediate after the patient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 190 | 264
Participants
  A lot of satisfaction | 149 | 193
  Some/Little Satisfaction | 30 | 58
  Missing/Unknown/No Discussion | 11 | 13

3. Primary Outcome: Communication Content
Description: PCP Explains CRC screening to my satisfaction
Time Frame: immediately after the patient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 190 | 264
Participants
  Strongly Agree | 152 | 203
  Somewhat Agree/Neither | 30 | 50
  Missing/Unknown/Did not Discuss | 8 | 11

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/190 | 1/264
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/264
Other Adverse Events (participants affected / at risk) | 0/190 | 0/264

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No